CLINICAL TRIAL: NCT03717493
Title: Deficits in Emotion Regulation Skills as a Maintaining Factor in Binge Eating Disorder
Acronym: ER-BED
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Friedrich-Alexander-Universität Erlangen-Nürnberg (Other)
Collaborators: German Research Foundation (Other); University of Freiburg (Other); University Hospital Tuebingen (Other)
Responsible Party: Principal Investigator, Matthias Berking, Ph.D., Head of department of clinical psychology, principle investigator, University of Erlangen-Nürnberg
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: BE4510/1-5
Record Dates: First submitted 2018-10-22; First posted 2018-10-24 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Binge-Eating Disorder
Keywords: Binge-Eating Disorder; Affect Regulation Training; Emotion Regulation; Transdiagnostic
MeSH Terms: conditions — Binge-Eating Disorder; Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial; group x time
Who Masked: Outcomes Assessor
Masking Description: Assessors were blinded with regard to study condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Affect Regulation Training (ART) (Experimental): Affect Regulation Training (ART; Berking & Whitley, 2014) is a transdiagnostic, group-based intervention aiming to enhance general affect regulation skills in individuals who meet criteria for mental disorders or are at-risk of developing mental-health problems.
  Interventions: Behavioral: Affect Regulation Training
- Waitlist Control Condition (WLC) (No Intervention): In order to control for the effects of time, we compared changes during ART with changes during WLC. Participants in the WLC condition received no treatment within the study but were offered to participate in ART after completing all assessments.

INTERVENTIONS:
Behavioral: Affect Regulation Training — Following the guidelines for the 6-week intensive ART format, we scheduled one 180-minutes session per week (each consisting of two modules à 90min) for a period of six subsequent weeks. Training groups included four to eight participants. The implementation of ART followed standardized treatment protocols (Berking & Whitley, 2014). ART was delivered by doctoral candidates (DCs) in clinical psychology who had completed or were in advanced stages of their clinical training. All therapists had been intensely trained and received weekly supervision from experienced ART trainers. To control adherence a random sample of 5% of all sessions was be videotaped and will be rated with regard to adherence.
  Arms: Affect Regulation Training (ART)

SUMMARY:
The effectiveness of a systematic affect regulation training (ART; Berking, 2010) is evaluated with regard to reducing symptoms of binge eating disoder in a randomized controlled trial.

DETAILED DESCRIPTION:
Evidence suggests that deficits in affect regulation play an important role in the development and maintenance of binge eating disorder (BED). Thus, we aim to clarify whether BED symptoms can be reduced with the help of a training of general affect regulation skills. For this purpose, we randomly allocated N = 99 individuals meeting criteria for BED either to an affect regulation training (ART) or to a wait list control condition (WLC). Primary outcome is the reduction of binges during the treatment-vs.-waiting period as assessed with the Eating Disorder Examination (EDE) interview. Secondary outcomes include BED symptom severity at follow-up and change in emotion regulation skills. To clarify whether potential differences between groups regarding change in binge eating result from a greater increase of affect regulation skills in ART, we will test whether potential group differences regarding binges will be mediated by differences between groups regarding change in affect regulation skills.

Change of randomization procedure: Over the course of the study, serious difficulties occurred with regard to recruiting participants as quickly as necessary to avoid drop-outs due to participants' unwillingness to wait until eight individuals were recruited for randomization. To solve the problem, we switched from the original block randomization to a procedure in which the next patient eligible for the study was allocated to the treatment condition until the minimum group size of four was reached.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of BED according to DSM-5 criteria
* age over 18 and below 69
* 25 < BMI < 45
* ability and willingness to provide informed consent

Exclusion Criteria:

* high risk of suicide
* co-occurring psychotic, bipolar disorders, alcohol/substance dependence within the past six months and/or borderline personality disorder
* medical disorders that would affect weight and/or the ability to participate
* insufficient German language skills (as assessments and treatment were conducted in German)
* current participation in psychotherapeutic treatment other than those offered in the study
* current participation in a weight control program
* taking medication that would affect weight
* pregnancy.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients were asked to report their gender.
Enrollment: 99 (Actual)
Dates: Start 2012-12-17 (Actual); Primary Completion 2017-05-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Number of binges | past 28 days
  Number of binges as assessed in the Eating Disorder Examination Interview (EDE; Fairburn & Cooper, 1993; German version: Hilbert & Tuschen-Caffier, 2006)

IPD SHARING:
Plan to Share IPD: Yes
Deidentified IPD will be made available upon request
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: From October 2018 to October 2028
Access Criteria: Credible reason for request